CLINICAL TRIAL: NCT00933322
Title: Randomized-controlled Trial to Assess the Effects of Different Trans-fatty Acids on Endothelial Function in Humans
Brief Title: Trial to Assess the Effects of Different Trans-fatty Acids on Endothelial Function in Humans
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment problems
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Agroscope Liebefeld-Posieux Research Station ALP (Other); University of Bern (Other); Schweizerische Herzstiftung (Other); Bundesamt für Landwirtschaft (Unknown); Emmi Schweiz AG (Unknown)
Responsible Party: Hugo Saner/ Prof. Dr. med, Bern University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: KEK 124/09
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Healthy
Keywords: ruminant; industrial; endothelial function; flow-mediated dilation; blood lipids; nutrition; trans fatty acids; coronary disease; endothelial function of the brachial artery; inflammation; insulin resistancy; coagulation
MeSH Terms: conditions — Coronary Disease; Inflammation; Thrombosis | interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ruminant TFA (Active Comparator): In addition to the basic diet, volunteers enrich their diet with an individually calculated amount of butter containing ruminant TFA and with 15-20g rape oil for balancing the essential fatty acids.
  Interventions: Dietary Supplement: diet enriched with ruminant trans fatty acids
- industrial TFA (Active Comparator): In addition to the basic diet, volunteers enrich their diet with an individually calculated amount of butter containing TFA from PHVO and with 15-20g rape oil for balancing the essential fatty acids.
  Interventions: Dietary Supplement: diet enriched with industrial trans fatty acids
- without TFA (Placebo Comparator): In addition to the basic diet, volunteers enrich their diet with an individually calculated amount of butter without TFA and with 15-20g rape oil for balancing the essential fatty acids.
  Interventions: Dietary Supplement: diet without any trans fatty acids

INTERVENTIONS:
Dietary Supplement: diet enriched with industrial trans fatty acids — After run-in phase of 2 weeks with margarine without TFA, 4 weeks with margarine enriched with industrial trans fatty acids following. TFA-percentage of total energy consumption is 2% or 6% of total fat energy consumption.
  Arms: industrial TFA
Dietary Supplement: diet enriched with ruminant trans fatty acids — After run-in phase of 2 weeks with margarine without TFA, 4 weeks with butter enriched with ruminant trans fatty acids following. TFA-percentage of total energy consumption is 2% or 6% of total fat energy consumption.
  Arms: ruminant TFA
Dietary Supplement: diet without any trans fatty acids — 6 weeks with margarine without any trans fatty acids.
  Arms: without TFA

SUMMARY:
The aim of the study is to compare a diet rich in trans fatty acids (TFA) from ruminant sources with a diet rich in TFA from hydrogenated vegetable oils (PHVO) in regard to their effects on cardiovascular risk markers (endothelial function, blood lipids, inflammation and coagulation parameters in the blood).

After a two week run-in period (diet without TFA) volunteers are randomized into three groups with different diets: diet rich in TFA from ruminant sources, diet rich in TFA from PHVO and diet without TFA. The intervention period lasts four weeks.

A nutritionist introduces the basic issues of the study diets. All volunteers supply themselves according to the recommendations of the Swiss food pyramid. Fat free food can be chosen individually in the context of defined guidelines. The amount and source of the fat in the diet are strictly defined. During the whole study, volunteers meet the nutritionist every 2 weeks, and in the weeks between, the volunteers are contacted by phone.

The volunteers will continue their normal daily life and physical activities. At the beginning of the run-in period and at the beginning and the end of the intervention period the endothelial function of the brachial artery will be assessed using flow-mediated dilation (FMD)/nitro-mediated dilation (NMD) methods and blood samples will be collected to analyze blood lipids, inflammation and coagulation parameters in the blood.

Hypothesis:

1. Diet enriched with ruminant TFA has not the same negative effect on cardiovascular risk markers as diet enriched with the same amount of industrial TFA compared with a diet without TFA.
2. Diet enriched with ruminant TFA has not a more negative effect on cardiovascular risk markers as diet without TFA.

DETAILED DESCRIPTION:
Background:

For some time already negative effects of trans fatty acids (TFA) on the cardiovascular system are known. The main TFA sources in our nutrition are partly hydrogenated vegetable oils (PHVO) which result from partially oil hardening.

TFA also occur naturally in ruminant fat (meat, milk and their products). Epidemiologic studies suggest that not all TFA have the same negative effects on the cardiovascular system.

As the detrimental effect of TFA from PHVO is unquestioned (Mozaffarian et al. 2006, Ascherio et al. 1999), TFA from ruminant origin may have a neutral or positive effect on the cardiovascular system (Pfeuffer und Schrezenmeir 2006, Willett et al. 1993). The main reason is attributed to the different concentrations of TFA-isomers in the fat depending on the origin. Partially hydrogenated vegetable oils contains a high amount of elaidic acids (trans-9 18:1 isomer) and trans-10 18:1 isomers. Ruminant fats contain a high amount of vaccenic acids (trans-11 18:1 isomer). The vaccenic acid can be converted to the harmless conjugated linoleic acid (CLA) in the human and ruminant metabolic system.

TFA from PHVO have a negative effect on blood lipids and markers of the inflammatory system. They increase the Low Density Lipoproteins (LDL) and decrease the High Density Lipoproteins (HDL). Markers of the inflammatory system as TNFa Receptors, IL-6 and CRP increase with TFA consumption (Mensink et al. 2003; Mozaffarian 2006; Mozaffarian et al. 2009).

The discussion on the effect of TFA on insulin sensitivity is discussed conversely since there exists few studies which show different results. The trend indicates an impairment of insulin sensitivity with TFA consumption, particularly in predisposed persons (Hu 2001; Mozaffarian 2009; Risérus 2006).

Other studies indicated a negative effect on vessels' endothelial function and increase the level of soluble adhesion molecules (ICAM, VCAM) which are markers of endothelial dysfunction (Mozaffarian 2006; Mozaffarian et al. 2006).

Almost every typical risk factors of cardiovascular diseases induce changes in endothelial function which can preclinically be detected.

The analysis of endothelial function using endothelium-dependent flow-mediated dilation (FMD)and endothelium-independent vasodilation with nitroglycerin (NMD) of the brachial artery is a valuable, non-invasive method to determine the influence of various factors on the endothelial function (Moens et al. 2005).

Since changes in periphery are consistent with changes in the coronary vessels (Anderson et al. 1995), FMD represent a valuable indicator for cardiac events (Gokce et al. 2002, 2003; Widlansky et al. 2003). FMD is defined as percentage increase in vessel diameter from baseline conditions to maximum vessel diameter during hyperaemia (de Roos et al. 2003a).

Previous comparisons between TFA from ruminants and PHVO in clinical studies were only focused on changes in blood lipids (Chardigny et al. 2008, Motard-Bélanger et al. 2008).

Blood lipids are important factors concerning the risk of cardiovascular diseases, but not the only one as epidemiological and clinical studies indicated.

Studies on the effect of TFA on endothelial function, as well as on inflammatory and coagulation markers in the blood, become more important.

Objective:

The aim of the study is to compare a diet rich in trans fatty acids (TFA) from ruminant sources with a diet rich in TFA from hydrogenated vegetable oils (PHVO) in regard to their effects on cardiovascular risk markers (endothelial function, blood lipids, inflammation and coagulation parameters in the blood).

Methods:

Randomized, controlled, double blind study with healthy volunteers of both sex, aged between 45-65y. About 200 volunteers will be enrolled and randomized into 3 parallel study arms after a run-in period of 2 weeks.

Group 1 will follow a diet with 2% TFA of the total energy consumption from ruminant source, group 2 a diet with 2E% TFA from PHVO and group 3 a diet without any TFA for 4 weeks.

At the beginning of the run-in period and at the beginning and the end of the intervention period the endothelial function of the brachial artery will be assessed using flow-mediated dilation (FMD)/ nitro-mediated dilation (NMD) methods and blood samples will be collected to analyse blood lipids, inflammation and coagulation parameters in the blood. Nutrition councils will be passed at the beginning of the run-in period and then every 2 weeks. In the weeks between, the volunteers are contacted by phone.

ELIGIBILITY:
Inclusion Criteria:

* age 45-69
* body mass index 20-30 kg/m2
* willingness to hold physical activity constant over study duration
* written informed consent

Exclusion Criteria

* smoking
* hypertension (> 140/90 mm Hg)
* hypotension (men < 115 mm Hg; women < 105 mm Hg)
* obesity (BMI =/> 30 kg/m2)
* vegan
* infections in the last 6 weeks
* allergy for food (e.g., milk)
* pregnancy
* diabetes (elevated fasting blood glucose level)
* clinical known coronary diseases
* acute and/or chronical medication (incl. contraceptive)
* abnormal kidney function
* abnormal liver function
* known cardiac arrhythmia (e.g., atrial fibrillation)
* blood parameters (ALAT, Creatinin, Hb, potassium, CRP) in range

Ages: 45 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2009-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
endothelial function using flow-mediated dilation | 3 time points over 6 weeks (after 0, 2, 6 weeks)

SECONDARY OUTCOMES:
inflammation parameters in blood samples | 6 weeks
coagulation parameters in blood samples | 6 weeks
blood lipids in blood samples | 6 weeks
adhesion molecules in blood samples | 6 weeks
insulin resistance via blood samples | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Saner, Prof. Dr. med, Study Director — Cardiovascular Prevention and Rehabilitation, University Hospital Bern, Switzerland; Alexandra Schmid, Dipl. oec. troph., Study Director — Agroscope Liebefeld-Posieux Research Station ALP, Posieux, Switzerland; Thomas Radtke, MSc, Principal Investigator — Cardiovascular Prevention and Rehabilitation, University Hospital Bern, Switzerland
Locations (1):
- Cardiovascular Prevention and Rehabilitation, Bern University Hospital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Background] Mozaffarian D, Katan MB, Ascherio A, Stampfer MJ, Willett WC. Trans fatty acids and cardiovascular disease. N Engl J Med. 2006 Apr 13;354(15):1601-13. doi: 10.1056/NEJMra054035. No abstract available. PMID 16611951
- [Background] Ascherio A, Katan MB, Zock PL, Stampfer MJ, Willett WC. Trans fatty acids and coronary heart disease. N Engl J Med. 1999 Jun 24;340(25):1994-8. doi: 10.1056/NEJM199906243402511. No abstract available. PMID 10379026
- [Background] Willett WC, Stampfer MJ, Manson JE, Colditz GA, Speizer FE, Rosner BA, Sampson LA, Hennekens CH. Intake of trans fatty acids and risk of coronary heart disease among women. Lancet. 1993 Mar 6;341(8845):581-5. doi: 10.1016/0140-6736(93)90350-p. PMID 8094827
- [Background] Moens AL, Goovaerts I, Claeys MJ, Vrints CJ. Flow-mediated vasodilation: a diagnostic instrument, or an experimental tool? Chest. 2005 Jun;127(6):2254-63. doi: 10.1378/chest.127.6.2254. PMID 15947345
- [Result] Mozaffarian D, Aro A, Willett WC. Health effects of trans-fatty acids: experimental and observational evidence. Eur J Clin Nutr. 2009 May;63 Suppl 2:S5-21. doi: 10.1038/sj.ejcn.1602973. PMID 19424218
- [Result] Chardigny JM, Destaillats F, Malpuech-Brugere C, Moulin J, Bauman DE, Lock AL, Barbano DM, Mensink RP, Bezelgues JB, Chaumont P, Combe N, Cristiani I, Joffre F, German JB, Dionisi F, Boirie Y, Sebedio JL. Do trans fatty acids from industrially produced sources and from natural sources have the same effect on cardiovascular disease risk factors in healthy subjects? Results of the trans Fatty Acids Collaboration (TRANSFACT) study. Am J Clin Nutr. 2008 Mar;87(3):558-66. doi: 10.1093/ajcn/87.3.558. PMID 18326592
- [Result] Motard-Belanger A, Charest A, Grenier G, Paquin P, Chouinard Y, Lemieux S, Couture P, Lamarche B. Study of the effect of trans fatty acids from ruminants on blood lipids and other risk factors for cardiovascular disease. Am J Clin Nutr. 2008 Mar;87(3):593-9. doi: 10.1093/ajcn/87.3.593. PMID 18326596
- [Derived] Guggisberg D, Burton-Pimentel KJ, Walther B, Badertscher R, Blaser C, Portmann R, Schmid A, Radtke T, Saner H, Fournier N, Butikofer U, Vergeres G. Molecular effects of the consumption of margarine and butter varying in trans fat composition: a parallel human intervention study. Lipids Health Dis. 2022 Aug 18;21(1):74. doi: 10.1186/s12944-022-01675-1. PMID 35982449
- [Derived] Radtke T, Schmid A, Trepp A, Dahler F, Coslovsky M, Eser P, Wilhelm M, Saner H. Short-term effects of trans fatty acids from ruminant and industrial sources on surrogate markers of cardiovascular risk in healthy men and women: A randomized, controlled, double-blind trial. Eur J Prev Cardiol. 2017 Mar;24(5):534-543. doi: 10.1177/2047487316680691. Epub 2016 Dec 5. PMID 27899529